CLINICAL TRIAL: NCT00022620
Title: Phase II Study On Paclitaxel In Recurrent Uterine Papillary Serous Carcinoma (UPSC)
Brief Title: Paclitaxel in Treating Patients With Refractory or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-55961; EORTC-55961
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Endometrial Cancer
Keywords: recurrent endometrial carcinoma; endometrial papillary serous carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients who have refractory or recurrent endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the therapeutic activity of paclitaxel in patients with refractory or recurrent endometrial papillary carcinoma.
* Determine the objective response and duration of response in patients treated with this regimen.
* Determine the acute side effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 12 weeks.

PROJECTED ACCRUAL: Approximately 16-29 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed endometrial papillary carcinoma (uterine papillary serous carcinoma)

  * Progressive or recurrent
* Bidimensionally measurable disease
* Platinum refractory disease, defined by one of the following:

  * Progression during platinum-based chemotherapy
  * Stable disease for at least 4 courses of platinum-based chemotherapy
  * Recurrence within 4 months of platinum-based chemotherapy
* No brain involvement or leptomeningeal disease

PATIENT CHARACTERISTICS:

Age:

* 75 and under

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 50 umol/L

Renal:

* BUN no greater than 8.0 mmol/L
* Creatinine no greater than 120 umol/L
* Creatinine clearance at least 60 mL/min

Other:

* Not pregnant
* Fertile patients must use effective contraception
* HIV negative
* No other prior or concurrent malignancy except basal cell carcinoma of the skin
* No active bacterial infection (e.g., urinary tract infection)
* No uncontrolled or potentially active site of infection (e.g., fistula or abscess)
* No psychological, familial, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* At least 1 prior platinum containing regimen
* At least 50 mg/m2 per course for a maximum of 28 days for cisplatin
* At least 5 times AUC for a maximum of 4 weeks per course for carboplatin
* Prior non-taxane-containing chemotherapy allowed

Endocrine therapy:

* At least 4 weeks since prior hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* At least 3 months since prior radiotherapy to target lesion
* Concurrent radiotherapy allowed for bone pain provided evaluable lesions are outside of irradiation field)

Surgery:

* Prior surgical management of lymph nodes allowed

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gitsch, MD, Study Chair — Allgemeines Krankenhaus - Universitatskliniken
Locations (8):
- Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Italy (2):
  - Ospedale Mauriziano Umberto I, Torino
  - Ospedale Civile, Voghera (PV)
- Hospitais da Universidade de Coimbra (HUC), Coimbra, Portugal
- Hospital Universitasrio San Carlos, Madrid, Spain
- Queen Elizabeth Hospital, Gateshead, England, United Kingdom